CLINICAL TRIAL: NCT00467701
Title: Prevalence of Legionella Infections, Bacterial Etiology in Pneumonia Among Patients Admitted to Hospital,- and Risk Factors/Characteristics for These Patients.(Translated From Norwegian)
Brief Title: Community Acquired Pneumonia in Telemark and Ostfold
Acronym: CAPITO
Status: Completed | Type: Observational
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: Sykehuset Ostfold (Other)
Responsible Party: Wenche Røysted, Sykehuset Telemark HF, Norway
Other Study IDs: STHF 5690.10; NSD: 16388; REK: S-05393
Record Dates: First submitted 2007-04-30; First posted 2007-05-01 (Estimated); Last update posted 2009-01-19 (Estimated); Status verified 2009-01

CONDITIONS: Community Acquired Pneumonia
Keywords: pneumonia; Legionnaires disease; risk factors
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia; Legionnaires' Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — sputum
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to investigate the bacterial causes in community acquired pneumonia in adults admitted to hospital in two counties in Norway and to look at possible factors that makes the patients susceptible to pneumonia.

DETAILED DESCRIPTION:
In Norway there is little knowledge of which bacterias that causes pneumonia in patients admitted to hospital. There are also few registered cases of Legionnaires disease every year, compared to our neighbour countries.

Therefore 500 patients with community acquired pneumonia admitted to Telemark hospital and Ostfold hospital in Norway will be tested by urin antigen test for the detection of Legionella pneumophila serogroup 1 and Streptococcus pneumoniae. We will also perform routine bacterial culture of sputum and culture on medium for isolation of Legionella species. A throat swab from the patients will be tested for Mycoplasma pneumoniae, Chlamydophila pneumoniae and Bordetella pertussis using PCR-techniques. Legionella-serology will also be performed. In addition all the included patients are invited to fill in a questionnaire in order to look for risk factors for developing community acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of lower airway infection and radiologic sings of pneumonia.

Exclusion Criteria:

* Age<18
* Serious psychiatric illness
* Mentally retarded
* Hospitalized last 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital with community acquired pneumonia.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Halfrid Waage, dr.med, Study Chair — Telemark Hospital, 3710 Skien, Norway
Locations (1):
- Sykehuset Telemark, Skien, Telemark, Norway